CLINICAL TRIAL: NCT01177358
Title: Botulinum Toxin A in the Healing of Surgical Wounds of the Neck: a Randomized, Prospective, Placebo-controlled Trial
Brief Title: Botox in the Healing of Surgical Wounds of the Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BTX-001
Record Dates: First submitted 2010-07-08; First posted 2010-08-09 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-10

CONDITIONS: Scar
Keywords: Scar; Botox
MeSH Terms: conditions — Cicatrix | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin A injection (Experimental): A vial of Botulinum Toxin A containing 100U of Botox will be reconstituted with 2mL of normal saline for a concentration of 50U/mL.
  5 Units (0.1 mL) of Botulinum Toxin A will be injected at three sites along the incision (midline and 1.5 cm lateral to midline) following a thyroidectomy or parathyroidectomy.
  Interventions: Drug: Botulinum Toxin Type A
- Saline (Placebo Comparator): 0.1 mL of normal saline in a placebo vial containing 2 mL of normal saline will be injected along the incision (midline and 1.5 cm lateral to midline) following a thyroidectomy or parathyroidectomy.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A — A vial of Botulinum Toxin A containing 100U of Botox will be reconstituted with 2mL of normal saline for a concentration of 50U/mL.
  5 units (0.1mL) of Botulinum Toxin a will be injected at midline and 1.5cm lateral to midline, bidirectionally, following a thyroidectomy or parathyroidectomy.
  Other Names: Allergan Botox; Drug Identification Number 01981501
  Arms: Botulinum Toxin A injection
Drug: Normal Saline — 0.1mL of normal saline in a placebo vial containing 2mL of normal saline will be injected along three sites (midline and 1.5cm lateral from midline) following a thyroidectomy or parathyroidectomy.
  Arms: Saline

SUMMARY:
The investigators hypothesize that Botox A will reduce scarring and improve healing of surgical neck wounds.

DETAILED DESCRIPTION:
Botulinum Toxin A is a toxin produced by the anaerobic bacterial species Clostridium botulinum. The toxin specifically inhibits release of the neurotransmitter Acetylcholine at synaptic junctions, thus preventing neuromuscular transmission, and inducing paralysis of the muscle.

Previous studies have indicated that tensile forces on the skin may affect the healing of a wound. These forces act against the immature collagen laid down during wound healing and may stimulate overgrowth, thereby contributing to the formation of hypertrophic scars or keloids.

Using botox to paralyse the underlying muscles may reduce the tensile force on the overlying skin, and thus reduce scar formation and promote healing. Botox has also been shown to affect the cell cycle distribution of fibroblasts derived from hypertrophic scars.

The objective of this study is to determine the effects of BTX-A in wound healing and the reduction of scar formation.

Patients undergoing a thyroidectomy or parathyroidectomy will be randomized to receive either BTX-A injections along the surgical site or placebo immediately following closure. All incisions will be sutured in a similar fashion. BTX-A or normal saline will then be injected along the platysma muscle. The patient and the surgeon will be blinded to the treatment arm. Photographs will be taken of the surgical site at 4 weeks and 6 months. The patient and two otolaryngologists will independently score the healing of the wound using a standardized scoring method. The scores be compared between the two surgeons to determine correspondence and interobserver reliability.

The scores of the two treatment arms will be compared to reveal the effect of BTX-A on wound healing.

ELIGIBILITY:
Inclusion Criteria:

* all patients referred to the ENT clinic for a thyroidectomy or parathyroidectomy

Exclusion Criteria:

* patients with missing information, including demographic information
* patients lost to follow up or have been followed for less than 6 months
* patients with known allergy to lidocaine
* patients in whom botox would be contraindicated in:
* known history of neuromuscular disorders (myasthenia gravis, amyotrophic lateral sclerosis, Eaton-Lambert syndrome)
* pregnant women
* known allergy to botox, albumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale | 6 months
  The surgeon will assess the healing of the surgical incision at 6 months and fill out the Vancouver Scar Scale following the operation.

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale | 4 weeks
  The surgeon and the patient will be asked to fill out the survey at 4 weeks following the operation.
Patient and Observer Scar Assessment Scale | 6 months
  The surgeon and the patient will be asked to fill out the survey at 6 months following the operation.
Vancouver Scar Scale | 4 weeks
  The surgeon will assess the healing of the surgical incision and fill out the Vancouver Scar Scale at 4 weeks following the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Taylor, FRCS, Principal Investigator — Capital District Health Authority Nova Scotia
Locations (1):
- Queen Elizabeth II Hospital, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Gassner HG, Sherris DA, Friedman O. Botulinum toxin-induced immobilization of lower facial wounds. Arch Facial Plast Surg. 2009 Mar-Apr;11(2):140-2. doi: 10.1001/archfacial.2009.3. No abstract available. PMID 19289689
- [Result] Gassner HG, Brissett AE, Otley CC, Boahene DK, Boggust AJ, Weaver AL, Sherris DA. Botulinum toxin to improve facial wound healing: A prospective, blinded, placebo-controlled study. Mayo Clin Proc. 2006 Aug;81(8):1023-8. doi: 10.4065/81.8.1023. PMID 16901024
- [Result] Wilson AM. Use of botulinum toxin type A to prevent widening of facial scars. Plast Reconstr Surg. 2006 May;117(6):1758-66; discussion 1767-8. doi: 10.1097/01.prs.0000209944.45949.d1. PMID 16651948
- [Result] Xiao Z, Zhang F, Cui Z. Treatment of hypertrophic scars with intralesional botulinum toxin type A injections: a preliminary report. Aesthetic Plast Surg. 2009 May;33(3):409-12. doi: 10.1007/s00266-009-9334-z. Epub 2009 Apr 9. PMID 19357910
- [Derived] Phillips TJ, Fung E, Rigby MH, Burke E, Hart RD, Trites JRB, Gassner HG, Taylor SM. The Use of Botulinum Toxin Type A in the Healing of Thyroidectomy Wounds: A Randomized, Prospective, Placebo-Controlled Study. Plast Reconstr Surg. 2019 Feb;143(2):375e-381e. doi: 10.1097/PRS.0000000000005264. PMID 30688903